CLINICAL TRIAL: NCT07320261
Title: Cardiac Computed Tomography Evaluation of Epicardial Adipose Tissue Differences Between Patients With Atrial Fibrillation and Non-Atrial Fibrillation Individuals
Brief Title: Cardiac CT Evaluation of EAT in AF vs. Non-AF Subjects
Acronym: CCT-EAT-AF-NA
Status: Not yet recruiting | Type: Observational
Sponsor: xiaoya wang (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Sponsor-Investigator, xiaoya wang, Associate Chief Physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: 2025-1638-1
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); CT
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Paroxysmal AF
- Persistent AF: Paroxysmal AF
- Sinus rhythm

SUMMARY:
The goal of this cross-sectional study is to explore the relationship between atrial structural characteristics (such as epicardial adipose tissue infiltration and atrial size) and atrial fibrillation (AF), as well as the differences in these characteristics among different AF subtypes. It will also clarify the independent association between pericardial fat distribution and AF (and its subtypes) after excluding confounding factors.

The main questions it aims to answer are:

* What are the differences in epicardial adipose tissue volume and atrial size among patients with sinus rhythm, paroxysmal AF, and persistent AF?
* Is pericardial fat distribution independently associated with AF and its subtypes after adjusting for confounding factors such as age, hypertension, and left atrial enlargement?

Researchers will enroll patients who undergo coronary CTA or left atrial CTA at The Second Affiliated Hospital of Zhejiang University School of Medicine, and match and divide them into three groups (sinus rhythm group, paroxysmal AF group, and persistent AF group) based on BMI and other factors. They will compare the differences in pericardial fat distribution and baseline characteristics among the three groups and analyze the independent association between pericardial fat and AF.

Participants will:

* Provide relevant clinical baseline data and CTA examination results
* Complete the collection of demographic information, medical history, and laboratory test data

The study duration is 6 months, starting from the date of ethical approval, with an expected end date of June 2026. A total of 600-900 participants (200-300 per group) will be enrolled to ensure the reliability and clinical applicability of the research conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo coronary CTA or left atrial CTA examination at The Second Affiliated Hospital of Zhejiang University School of Medicine;
* Aged 18 years or older
* Cardiac rhythm status is confirmed as sinus rhythm, paroxysmal atrial fibrillation, or persistent atrial fibrillation;
* Willing to provide clinical baseline data and allow access to CTA examination results;
* Able to understand and cooperate with the data collection process of the study.

Exclusion Criteria:

* Patients with incomplete clinical baseline data or unreadable CTA images;
* Aged less than 18 years
* Patients who refuse to participate in the study or cannot cooperate with data collection;
* Other situations judged by the researchers to be unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older who undergo coronary CTA or left atrial CTA examination at The Second Affiliated Hospital of Zhejiang University School of Medicine. Participants will be categorized into three cohorts according to their confirmed cardiac rhythm status: sinus rhythm, paroxysmal atrial fibrillation, or persistent atrial fibrillation. All enrolled individuals must be willing to provide clinical baseline data and allow access to their CTA examination results, and be able to understand and cooperate with the study's data collection process. Patients under 18 years of age, those with incomplete clinical data or unreadable CTA images, and those who refuse to participate or cannot cooperate will be excluded from the study. The total planned sample size is 600-900 participants, with 200-300 participants in each cohort.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The difference in epicardial adipose tissue distribution among the three cohorts | At the time of enrollment

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers upon reasonable request. The shared data will include de-identified participant information relevant to the study objectives, such as demographic data, clinical baseline characteristics, CTA examination results, and statistical analysis datasets. To protect participant privacy, all shared data will be de-identified by removing personal identifiers (e.g., name, ID number, contact information) in accordance with ethical regulations and data protection policies of The Second Affiliated Hospital of Zhejiang University School of Medicine. Researchers requesting IPD must submit a research proposal demonstrating the scientific relevance of their study, agree to abide by data use agreements, and ensure that the shared data is only used for legitimate scientific research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will be initiated after the primary study results are published, and the sharing period will be 3 years from the date of publication.
Access Criteria: Researchers engaged in legitimate scientific research related to the study field (e.g., cardiovascular disease research focusing on atrial fibrillation and atrial structural characteristics) who can demonstrate the scientific relevance and feasibility of their research projects.
  De-identified IPD and supporting information including the study protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) template, Clinical Study Report (CSR), and analytic code.
  How to access: Interested researchers should first submit a formal application to the research team of The Second Affiliated Hospital of Zhejiang University School of Medicine, which includes a detailed research proposal, proof of institutional affiliation, and a commitment to abide by relevant ethical regulations and data use agreements. After the research team reviews and approves the application, the de-identified IPD and supporting information will be provided.